CLINICAL TRIAL: NCT05775302
Title: Effects of Instrument-Assisted Soft Tissue Mobilization on Gastrocnemius and Achilles Tendon in Plantar Fasciitis
Brief Title: Instrument-Assisted Soft Tissue Mobilization on Gastrocnemius and Achilles Tendon in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Parwasha Shoukat
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Plantar Fascitis
Keywords: plantar Fascitis; Ache; Joint Range of Motion; Disability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM Gastrocnemius (Experimental): Instrument assisted soft tissue mobilization on gastrocnemius
  Conventional therapy:
  Cryotherapy for 10 min stretching of calf and plantar fascia strengthning of intrinsic foot muscle
  Interventions: Other: IASTM of Gastrocnemius + Conventional therapy
- IASTM Achillies Tendon (Active Comparator): Instrument assisted soft tissue mobilization Achillies Tendon
  Conventional therapy:
  Cryotherapy for 10 min stretching of calf and plantar fascia strengthning of intrinsic foot muscle
  Interventions: Other: IASTM of AchillesTendon + Conventional Therapy

INTERVENTIONS:
Other: IASTM of Gastrocnemius + Conventional therapy — The SWEEP technique will be performed downwards from the popliteal region to the Achilles tendon for 60 seconds, 30 times 12 sessions over a time frame of 4 weeks at a frequency of 3 sessions per week.
  Arms: IASTM Gastrocnemius
Other: IASTM of AchillesTendon + Conventional Therapy — Participants will receive a maximum of 60 seconds<30 times 12 sessions over a time frame of 4 weeks at a frequency of 3 sessions per week.
  Arms: IASTM Achillies Tendon

SUMMARY:
Aim of this study is to compare the effects of instrument assisted soft tissue mobilization on gastrocnemius and Achilles tendon on pain,range of motion and foot disability.A randomized control trial that will include total 32 participants and divided into two groups.Patients in Group A will receive instrument assisted soft tissue mobilization of gastrocnemius and Group B will receive instrument assisted soft tissue mobilization of Achilles tendon. While conventional therapy will be given to both groups.Data collected will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Plantar fasciitis is typical condition that produces pain in the medial longitudinal arch of the foot.Repetitive traction stresses on the plantar fascia at its origin over the distal calcaneus obesity, the makeup of the feet, and lifestyle choices are all factors that might contribute to the development of PF.

Physiotherapy interventions includes stretching the gastrocnemius and soleus,dry needling, IASTM (instrument assisted soft tissue mobilisation), exercise therapy, ultrasound therapy, iontophoresis, laser therapy, splints, and taping.Use of Instrument-Assisted Soft Tissue Massage has increased in popularity, and the plantar fascia is a superficial tissue that may benefit from this treatment.The Graston Technique Instrument-assisted Soft Tissue Mobilisation not only increases blood flow and tissue healing to the area as well as breaking up soft tissue restrictions along with increase fibroblasts, mast cell production and phagocytes.

Previous literature were limited in sample size, and only immediate effects of these techniques were studied But this study opted for the long term use of graston technique on gastrocnemius in comparison on Achilles tendon. So the purpose of this study is to compare the effects of Graston technique instrument assisted soft tissue mobilization at gastrocnemius and Achilles tendon in patients with planter fascitis. It will add to the growing body of knowledge that if same technique on different soft tissues will yield comparable outcomes,which should be the alternate choice of therapy

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Participants between age of 25 and 50 years
* Patients with maximal pain located at the antero-medial aspect of the plantar surface of the calcaneus
* Pain aggravated by passive dorsiflexion or standing/ walking on the big toe
* Patients with pain on taking first step in the morning(18)
* Patient volunteer to participate in the study and signed informed consent.

Exclusion Criteria:

* Patient with history of musculoskeletal disorders.
* Patient with any previous history of ankle or foot surgery.
* Patient with history of ankle or foot fracture.
* Patient with severe bone disorder (osteoporosis)
* Patient with history of Venous insufficiency.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Visual analogue scale id used to measures pain intensity. It consists of a 10cm line, with two end points representing 0 ('no pain') and 10 (pain as bad as it could possibly be)

SECONDARY OUTCOMES:
Goniometer | 4 weeks
  Goniometer is used to measure the ROM of joints
Foot and ankle disability index | 4 weeks
  Foot and Ankle Disability Index is a 34-item questionnaire divided into two subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MSOMPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Adam Life Care, Rawalpindi, Punjab Province
  - Attock Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No